CLINICAL TRIAL: NCT03488758
Title: Enjoyment of Infant Formulas Based on Cow or Goat Milk Protein
Acronym: CHARLIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHARLIE
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Feeding Behavior; Feeding, Bottle
MeSH Terms: conditions — Feeding Behavior; Bottle Feeding | interventions — Glia Maturation Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMF (Active Comparator): infant formula based on cow milk protein fractions
  Interventions: Other: CMF
- GMF (Experimental): infant formula based on whole goat milk
  Interventions: Other: GMF

INTERVENTIONS:
Other: CMF — Taking a infant formula based on cow milk protein fractions, 4-5 feeds per day given by bottle, 180-210 ml/feed, total 800-900ml per day for one mounth
  Arms: CMF
Other: GMF — Taking a infant formula based on whole goat milk, 4-5 feeds per day given by bottle, 180-210 ml/feed, total 800-900ml per day for one mounth
  Arms: GMF

SUMMARY:
To assess parental perceptions on infant feeding behavior and enjoyment with a goat milk formula compared to a cow milk formula

DETAILED DESCRIPTION:
This is a feasibility study to determine the utility of two new standardized psychometric tools for paediatricians to assess and manage feeding difficulties in formula fed infants. Baby Eating Behaviour Questionnaire (BEBQ) and Montreal Children's Hospital Feeding Scale (MCH-Feeding Scale) will be used in this study.

The secondary objectives are to determine if these tools can then measure the changes in behaviour after introducing two formula that differ in the sources of protein, ie formula made from whole goat milk compared to a conventional formula made from cow milk proteins. The quality of life and general health outcomes of these infants will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 2-3 months, predominantly formula fed

Exclusion Criteria:

* Infants born less than 37GA
* Confirmed or suspected cow milk protein allergy
* Predominantly breast fed
* Infants suffering from chronic disease

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Feeding enjoyment score from Baby Eating Behaviour Questionnaire (BEBQ). | 1 month
  Feeding enjoyment score from Baby Eating Behaviour Questionnaire (BEBQ).

SECONDARY OUTCOMES:
Feeding behaviour assessed by Montreal Children's Hospital Feeding Scale | 1 month
  This feeding scale permit to distinguish babies with no feeding difficulties (score under 61) or with mild (61-65) , moderate (65-70), or severe feeding disorders (>70)
Quality of life assessed by QUALIN | 1 month
  Quality of life assessed by QUALIN
Formula liking, using 4-point visual analog scale (VAS) | 1 month
  Formula liking, using 4-point visual analog scale (VAS). The range of this scale goes from 0 (my baby hates this fomula) to 10 (my baby loves this formula)
Incidences of rash | 1 month
  Incidences of rash
Incidences of dry skin | 1 month
  Incidences of dry skin
Incidences of eczema | 1 month
  Incidences of eczema
Gastrointestinal symptoms | 1 month
  Gastrointestinal symptoms
Weight | 1 month
Height | 1 month
head circomference | 1 month

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - 2 Avenue Camille Blanc,, Beausoleil
  - 20 avenue du général Sarail, Chatou
  - 65 Avenue Henri Barbusse,, Le Blanc-Mesnil
  - 53 Boulevard De La Liberté, Les Lilas
  - 41 Rue Aristide Briand,, Levallois-Perret
  - 157 Avenue du Général Leclerc, Maisons-Alfort
  - 169 Avenue Achille Peretti, Neuilly-sur-Seine
  - 4 Rue Edouard Quenu, Paris
  - 67 Rue Condorcet,, Paris
  - 67 Rue Condorcet, Paris
  - 92 Avenue de la République, Paris
  - CHU Robert Debré, 48 Bd Sérurier, Paris
  - 3 Allée du 8 Mai 1945,, Suresnes
  - 13 Villa Beauséjour, Vincennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrosoli R, Di Stasio L, Mazzocco P. Content of alpha S1-casein and coagulation properties in goat milk. J Dairy Sci. 1988 Jan;71(1):24-8. doi: 10.3168/jds.S0022-0302(88)79520-X. PMID 3372804
- [Background] Bates JE, Freeland CA, Lounsbury ML. Measurement of infant difficultness. Child Dev. 1979 Sep;50(3):794-803. PMID 498854
- [Background] Berseth CL, Mitmesser SH, Ziegler EE, Marunycz JD, Vanderhoof J. Tolerance of a standard intact protein formula versus a partially hydrolyzed formula in healthy, term infants. Nutr J. 2009 Jun 19;8:27. doi: 10.1186/1475-2891-8-27. PMID 19545360
- [Background] Forsyth BW, McCarthy PL, Leventhal JM. Problems of early infancy, formula changes, and mothers' beliefs about their infants. J Pediatr. 1985 Jun;106(6):1012-7. doi: 10.1016/s0022-3476(85)80260-2. PMID 3998939
- [Background] Iacono G, Merolla R, D'Amico D, Bonci E, Cavataio F, Di Prima L, Scalici C, Indinnimeo L, Averna MR, Carroccio A; Paediatric Study Group on Gastrointestinal Symptoms in Infancy. Gastrointestinal symptoms in infancy: a population-based prospective study. Dig Liver Dis. 2005 Jun;37(6):432-8. doi: 10.1016/j.dld.2005.01.009. Epub 2005 Mar 2. PMID 15893282
- [Background] Infante DD, Segarra OO, Redecillas SS, Alvarez MM, Miserachs MM. Modification of stool's water content in constipated infants: management with an adapted infant formula. Nutr J. 2011 May 19;10:55. doi: 10.1186/1475-2891-10-55. PMID 21595890
- [Background] Kunz C, Lonnerdal B. Human-milk proteins: analysis of casein and casein subunits by anion-exchange chromatography, gel electrophoresis, and specific staining methods. Am J Clin Nutr. 1990 Jan;51(1):37-46. doi: 10.1093/ajcn/51.1.37. PMID 1688683
- [Background] Llewellyn CH, van Jaarsveld CH, Johnson L, Carnell S, Wardle J. Development and factor structure of the Baby Eating Behaviour Questionnaire in the Gemini birth cohort. Appetite. 2011 Oct;57(2):388-96. doi: 10.1016/j.appet.2011.05.324. Epub 2011 Jun 6. PMID 21672566
- [Background] Long T, Johnson M. Living and coping with excessive infantile crying. J Adv Nurs. 2001 Apr;34(2):155-62. doi: 10.1046/j.1365-2648.2001.01740.x. PMID 11430276
- [Background] Manificat S, Dazord A, Langue J, Danjou G, Bauche P, Bovet F, Cubells J, Luchelli R, Tockert E, Conway K. [Evaluation of the quality of life of infants and very young children: validation of a questionnaire. Multicenter European study]. Arch Pediatr. 2000 Jun;7(6):605-14. doi: 10.1016/s0929-693x(00)80127-x. French. PMID 10911526
- [Background] Mitchell DJ, McClure BG, Tubman TR. Simultaneous monitoring of gastric and oesophageal pH reveals limitations of conventional oesophageal pH monitoring in milk fed infants. Arch Dis Child. 2001 Mar;84(3):273-6. doi: 10.1136/adc.84.3.273. PMID 11207184
- [Background] Nowacki J, Lee HC, Lien R, Cheng SW, Li ST, Yao M, Northington R, Jan I, Mutungi G. Stool fatty acid soaps, stool consistency and gastrointestinal tolerance in term infants fed infant formulas containing high sn-2 palmitate with or without oligofructose: a double-blind, randomized clinical trial. Nutr J. 2014 Nov 5;13:105. doi: 10.1186/1475-2891-13-105. PMID 25373935
- [Background] Polack FP, Khan N, Maisels MJ. Changing partners: the dance of infant formula changes. Clin Pediatr (Phila). 1999 Dec;38(12):703-8. doi: 10.1177/000992289903801202. PMID 10618762
- [Background] Ramsay M, Martel C, Porporino M, Zygmuntowicz C. The Montreal Children's Hospital Feeding Scale: A brief bilingual screening tool for identifying feeding problems. Paediatr Child Health. 2011 Mar;16(3):147-e17. doi: 10.1093/pch/16.3.147. PMID 22379377
- [Background] Recio I, Perez-Rodriguez ML, Amigo L, Ramos M. Study of the polymorphism of caprine milk caseins by capillary electrophoresis. J Dairy Res. 1997 Nov;64(4):515-23. doi: 10.1017/s0022029997002343. PMID 9403766
- [Background] Savino F, Cresi F, Maccario S, Cavallo F, Dalmasso P, Fanaro S, Oggero R, Vigi V, Silvestro L. "Minor" feeding problems during the first months of life: effect of a partially hydrolysed milk formula containing fructo- and galacto-oligosaccharides. Acta Paediatr Suppl. 2003 Sep;91(441):86-90. doi: 10.1111/j.1651-2227.2003.tb00653.x. PMID 14599049
- [Background] Zhou SJ, Sullivan T, Gibson RA, Lonnerdal B, Prosser CG, Lowry DJ, Makrides M. Nutritional adequacy of goat milk infant formulas for term infants: a double-blind randomised controlled trial. Br J Nutr. 2014 May;111(9):1641-51. doi: 10.1017/S0007114513004212. Epub 2014 Feb 6. PMID 24502951
- [Derived] Jung C, Gonzalez Serrano A, Batard C, Seror E, Gelwane G, Poidvin A, Lavallee I, Elbez A, Brussieux M, Prosser C, Gallier S, Bellaiche M. Whole Goat Milk-Based Formula versus Whey-Based Cow Milk Formula: What Formula Do Infants Enjoy More?-A Feasibility, Double-Blind, Randomized Controlled Trial. Nutrients. 2023 Sep 19;15(18):4057. doi: 10.3390/nu15184057. PMID 37764840